CLINICAL TRIAL: NCT06112522
Title: Open, Prospective Study Evaluating the Efficacy and Safety of 0.05% Tirbanubulin (Klisiry®) in the Treatment of Basal Cell Carcinoma
Brief Title: Tirbanubulin (Klisiry®) in the Treatment of Basal Cell Carcinoma
Acronym: Tirbaso
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-PP-04
Record Dates: First submitted 2023-10-13; First posted 2023-11-01 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Cell Carcinoma
Keywords: TIRBANIBULIN
MeSH Terms: interventions — tirbanibulin

STUDY DESIGN:
Intervention Model Description: Single-Arm, Open-Label, Single Center
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental : 5 Day treatment course 1 with Tirbanibulin Ointment 1% (Experimental): Subjects will be given one study kit containing single-dose packets of Tirbanibulin Ointment 1% and instructed to topically apply to the treatment area once daily for 5 consecutive days. Subjects with unresolved lesion at d28 or d56 or d72 or d84 will be given an additional study kit containing single-dose packets of Tirbanibulin Ointment 1% and instructed to topically apply to the treatment area once daily for 5 consecutive days.
  Interventions: Drug: Tirbanibulin

INTERVENTIONS:
Drug: Tirbanibulin — Subjects will be given one study kit containing single-dose packets of Tirbanibulin Ointment 1% and instructed to topically apply to the treatment area once daily for 5 consecutive days. Subjects with unresolved lesion at d28 or d56 or d72 or d84 will be given an additional study kit containing single-dose packets of Tirbanibulin Ointment 1% and instructed to topically apply to the treatment area once daily for 5 consecutive days.
  Other Names: Tirbaso

SUMMARY:
his is a Phase 2, Single-Arm, Open-Label, Single Center, to Assess Efficacy and Safety of Tirbanibulin Ointment 1% in Adult Subjects with superficial basal cell carcinoma (sBCC) not arising on the face or scalp

DETAILED DESCRIPTION:
This is a pilot study aimed at studying the efficacy and tolerance of a new topical treatment regimen in BCC. The number of 50 sBCC to be treated was established based on previous studies that have investigated the effectiveness of a topical regimen in sBCC. Considering that approximately 10% of BCCs will be wrongly included or not evaluable or will present with a deviation protocol major, a total of 55 sBCC will be included in the study.Inclusion Criteria :

* Age > 18 years
* Histologically confirmed, primary, previously untreated, superficial basal cell carcinoma (sBCC) not arising on the face or scalp, ≤ 15 mm (large axis)

Exclusion Criteria :

* BCC of the face or scalp
* BCC of non-superficial subtype
* BCC with large axis > 15mm
* Relapsing BCC
* Allergy to treatment
* Treatment with cryotherapy, imiquimod, PDT, or radiotherapy in the BCC area during the 6 months prior to the screening visit. Visits : 1) Selection visit = V0: if the patient meets the selection criteria, oral and written information will be given to him. If the patient signs the consent during this consultation, the inclusion visit will be carried out at the same time. 2) Inclusion visit and start of treatment = V1 (D1): for patients who have not signed their consent at the previous visit, consent will be collected • Verification of inclusion and non-inclusion criteria • Collection of medical and surgical history • Collection of previous and concomitant treatments • Clinical evaluation by visual inspection: measurement of the long axis, calculation of the surface to be treated (maximum treated surface for all sBCC should not exceed > 25 cm2) • Realization of a layer with the limits of the lesion • Clinical photos • Examination by LC-OCT • Dispensing of Tirbanibulin for the treatment cycle (1 tube for up to 3 sBCC) • Explanation of the mode of application to the patient • First application performed on site • Giving the patient a notebook to record the applications of the product and local skin reactions. 3) Follow-up visit +/- retreatment = V2 (D28 ± 2 d) • Collection of adverse events and changes in concomitant treatments • Collection of local skin reactions in the patient notebook • Evaluation of local skin reactions • Clinical evaluation and by LC-OCT -> In case of cure clinically and by LC-OCT (complete remission, CR) end of the study for the patient -> In the absence of CR processing as in V1 -> in case of a wound at the application site, the study will end for the patient and he will be treated according to standard recommendantions for• sBCC 4) Additional follow-up visits +/- retreatment = V3 (D56±2 days), V4 (D84+/-2d) : these visits will be conducted identically to V2. 5) Short-term efficacy visit = V5 (D112 +/- 2d): same as V2 w/o treatment with Tirbanibulin. Patients not in CR will terminate the study and will be treated according to standard recommendations for sBCC. 6) Long-term efficacy visit = V6 (M12): same as V2 w/o treatment with Tirbanibulin. All patients will terminate the study. Patients with relapse of their BCC will be treated according to standard recommendations for sBCC.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Histologically confirmed,
* primary, previously untreated,
* superficial basal cell carcinoma (sBCC) not arising on the face or scalp, ≤ 15 mm (large axis)

Exclusion Criteria:

* BCC of the face or scalp
* BCC of non-superficial subtype
* BCC with large axis > 15mm
* Relapsing BCC
* Allergy to treatment
* Treatment with cryotherapy, imiquimod, PDT, or radiotherapy in the BCC area during the 6 months prior to the screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | up to 17 months
  IMC

SECONDARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | up to 17 months
  Type, frequency, severity and time to onset of adverse effects. Adverse effects will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) scale. Local adverse effects will be assessed by the LSR score.
Number of Participants With complete remission | After the treatment at 17 months
  Complete remission after the 1st, 2nd, 3rd or 4th cycle of Tirbanibulin (Klisiry®) in sBCC.
Number of participants with sBCC thickness. | Baseline visit
  sBCC thickness assessed

CONTACTS AND LOCATIONS:
Overall Officials: philippe Bahadoran, PhD, Principal Investigator — CHU de Nice, Service de Dermatologie
Locations (1):
- CHU de Nice - Hôpital de l'Archet, Nice, Alpes-maritimes, France

IPD SHARING:
Plan to Share IPD: No